CLINICAL TRIAL: NCT04857905
Title: Dose-staged Gamma Knife Radiosurgery Versus Microsurgical Resection - Evaluation of Neurosurgical Treatment Methods for Patients With Larger Brain Metastases - an Explorative Prospective Study
Brief Title: Dose-staged Gamma Knife Radiosurgery Versus Microsurgical Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Josa M Frischer, MD, PhD, Principal Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK 1623/2020
Record Dates: First submitted 2021-04-15; First posted 2021-04-23 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Brain Metastases
Keywords: Gamma Knife Radiosurgery; Brain metastases; Microsurgical resection
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microsurgical Resection of larger Brain Metastasis (Other): Patients over 18 years and under 90 years Patients with KPS ≥70 Patients with NSCLC, melanoma, breast cancer or renal cancer as primary tumor Maximum of three brain metastases on the diagnostic MRI Tumor volume of 8-20 ccm3 on the diagnostic MRI Lobular brain metastases Patients without any contraindications for both treatment options Written, signed informed consent for study particaption after counseling
  -> Patients who after counseling decide for microsurgical resection of their brain metastasis
  Interventions: Procedure: Microsurgical resection
- Radiosurgery of larger Brain Metastasis (Other): Patients over 18 years and under 90 years Patients with KPS ≥70 Patients with NSCLC, melanoma, breast cancer or renal cancer as primary tumor Maximum of three brain metastases on the diagnostic MRI Tumor volume of 8-20 ccm3 on the diagnostic MRI Lobular brain metastases Patients without any contraindications for both treatment options Written, signed informed consent for study particaption after study counseling
  -> Patients who after counseling decide for dose-staged radiosurgical treatment of their brain metastasis
  Interventions: Procedure: Gamma Knife radiosurgery

INTERVENTIONS:
Procedure: Microsurgical resection — Depending on the patient's choice, the microsurgical resection of the brain metastases will be performed.
  Arms: Microsurgical Resection of larger Brain Metastasis
Procedure: Gamma Knife radiosurgery — Depending on the patient's choice, the radiosurgical treatment of the brain metastases will be performed.
  Arms: Radiosurgery of larger Brain Metastasis

SUMMARY:
Background. Brain metastases (BM) are the most common intracranial tumor and occur in 20-40% of all oncological patients. The most common primary cancer in brain metastases is lung cancer, followed by melanoma, breast cancer, renal cancer and colorectal cancer. The incidence of brain metastases has been increasing but the occurrence of brain metastases is still associated with high morbidity and poor prognosis. The main treatment methods are stereotactic radiosurgery (SRS), microsurgical resection and whole brain irradiation (WBRT). In contrast to microsurgical resection, Gamma Knife radiosurgery (GKRS) is a non-invasive neurosurgical method, which allows treatment in multimorbid patients with contraindications for surgery in general anesthesia. Furthermore, stereotactic radiosurgery is the only local treatment method for multiple disseminated and thereby non-resectable brain metastases. In general, microsurgical resection is considered the treatment of choice for BM exceeding >3 cm in diameter. However, since the establishment of the dose-staged technique, larger metastases can also be treated radiosurgically in selected patients. This novel method allows the application of high cumulative dose for the treatment of complex brain metastases.

Aim. The aim of the study is to evaluate the clinical outcome in brain metastases patients with tumor volume between 8 and 20 ccm3. The clinical outcome will be compared between surgically and radiosurgically treated BM patients.

Patients and methods. The investigators plan to conduct an explorative prospective study including about 50 radiosurgically and 50 surgically treated patients with brain metastases. If a patient fulfill study-relevant inclusion criteria at the time of BM diagnosis, the principle study investigator will offer both treatment options to the patient. Depending on patient's choice, he/she will be categorized either to surgical or to radiosurgical treatment group. For the outcome evaluation of the different treatment options, a comprehensive database will be established. The study participations will not interfere with any clincally indicated therapeutic decisions and the study participants will not be exposed to any additional risks since both treatments represent suitable therapy options.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years and under 90 years
* Patients with KPS ≥70
* Patients with NSCLC, melanoma, breast cancer or renal cancer as primary tumor
* Maximum of three brain metastases on the diagnostic MRI
* Tumor volume of 8-20 ccm3 on the diagnostic MRI
* Lobular brain metastases
* Patients without any contraindications for both treatment options
* Written, signed informed consent for study particaption after study explanation

Exclusion Criteria:

* Patients under 18 years and over 90 years
* Patients with KPS <70
* Patients with other primary tumor
* More than three brain metastases on the diagnostic MRI
* Tumor volume <8 or >20 ccm3 on the diagnostic MRI
* Patients with contraindications for both treatment options

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Through completion of the study, an average of 1 year
  Time from first treatment

SECONDARY OUTCOMES:
Local tumor progression | Through completion of the study, an average of half a year
  Time from first treatment until local tumor progression

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No